CLINICAL TRIAL: NCT03431779
Title: Adipose Derived Stem Cell Transplantation Via Lipofilling for Vestibulodynia: a Controlled Intervention Study
Brief Title: Lipofilling as a Treatment for Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-01060
Record Dates: First submitted 2018-01-25; First posted 2018-02-13 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Vestibulodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Intervention Model Description: However, subjects in the lipofilling group will be able to undergo surgery (excision) 3 months after the lipofilling of this intervention did not have the requested effect.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adipose derived stem cell transplantation via lipofilling (Experimental): Liposuction of 60cc abdominal fat with its adipose derived stem cells which will be reinjected (10-20 cc) in the vestibular area after centrifugation for 3 minutes at 1000 rpm and decantation of oil and red blood cells.
  Interventions: Procedure: Adipose derived stem cell transplantation via lipofilling
- Surgical excision (Active Comparator): Excision of painful areas
  Interventions: Procedure: Surgical excision

INTERVENTIONS:
Procedure: Adipose derived stem cell transplantation via lipofilling — Liposuction of 60cc abdominal fat with its adipose derived stem cells which will be reinjected (10-20 cc) in the vestibular area after centrifugation for 3 minutes at 1000 rpm and decantation of oil and red blood cells.
  Arms: Adipose derived stem cell transplantation via lipofilling
Procedure: Surgical excision — Excision of painful areas
  Arms: Surgical excision

SUMMARY:
The investigators would like to investigate if lipofilling with its adipose derived stem cells (ADSC) could be a new, less invasive but equally or more effective therapeutic option for women with vestibulodynia than vestibulectomy. The investigators expect the study to be successful because of the anti-inflammatory effects of the ADSC and its effectiveness -although not thoroughly studied- in some neuropathic pain disorder like pudendal neuralgia or post mastectomy pain syndrome.

Method: A controlled intervention study: one group receiving golden standard therapy 'vestibulectomy' and one group receiving vestibular lipofilling.

ELIGIBILITY:
Inclusion Criteria:

* Vestibulodynia requesting surgery

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female subjects can be included.
Enrollment: 9 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Q-tip scores (Cotton swab assessment of vaginal pain) 3 months after surgery | 3 months after surgery
  Very light pressure along specific points in the area of the vulvar vestibule and where there is tenderness, asking the patient to characterize the tenderness on a scale of 0-10, whether it's no pain or exquisite pain and then plotting that on a diagram. Most physicians will find that in women with vestibulitis, the tenderness is most pronounced just below the hymenal margin and around the orifices of the so-called "Bartholin" gland ducts.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No